CLINICAL TRIAL: NCT02692950
Title: Perceptions of Advance Directive Formats-A Pilot Study
Brief Title: Patient Perception of Video Advance Care Planning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Paul S. Mueller, MD, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 15-008704
Record Dates: First submitted 2016-02-23; First posted 2016-02-26 (Estimated); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Advanced Directive Planning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dialysis Patients (Other): Honor My Decisions Advance Care Planning Videos, self-recorded by a patient using a computer application, followed immediately by a post-video questionnaire and a follow-up questionnaire 2-4 weeks later.
  Interventions: Other: Honor My Decisions Advance Care Planning Video; Behavioral: Post-video questionnaire

INTERVENTIONS:
Other: Honor My Decisions Advance Care Planning Video — Honor My Decisions is a commercial computer application which allows a person to record a video of his/her advanced care planning and legacy information.
Behavioral: Post-video questionnaire — Questions regarding the video process, changes to previous answers and reaction received by others viewing the video

SUMMARY:
Rates of advance directive completion among Americans, even those suffering from serious chronic illness, are notoriously poor. Moreover, the contents of completed advance directives are often difficult to interpret in the face of a medical crisis. The study aims to examine patient perceptions of electronic, interactive versions of advance care planning documentation.

DETAILED DESCRIPTION:
The investigators are studying the video platform of a commercially available advance directive application, Honor My Decisions. This application was generated with funding from patient advocacy groups. The application allows a person to create a legally valid advance directive on his or her own tablet or smart phone and share that directive (either by printing or emailing a secure link to family and/or health care providers). Additionally, the app includes a feature by which individuals may record several 2-4 minute videos to memorialize their health preferences, and also to leave a more personal message for loved ones (a video legacy).

The research team has compiled a list of question prompts for these advance care planning videos with the assistance of a panel of experts on communication, palliative care, critical care, ethics and the law. The investigators collected prompt suggestions from these 9 experts with a modified Delphi technique, using iterative surveys to generate consensus. The experts were instructed to consider both contents and phrasing of question prompts, to promote usability and also later utility (if the patient later became unable to speak for him- or herself). These question prompts will form the basis of this pilot study.

The investigators aim to assess the experiences of patients completing electronic advance directives and documenting their care preferences and personal legacy via video. Renal dialysis patients have been selected as a patient population with frequent hospitalizations and low rates of advance directive completion. Patients will be given the opportunity to interact with the application and record their own videos. They will then provide immediate and long-term feedback about the video question prompts via interview.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing dialysis treatment
* 18 years of age or older

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-02; Primary Completion 2016-06-05 (Actual); Study Completion 2016-06-05 (Actual)

PRIMARY OUTCOMES:
Number of advanced care planning videos completed | Approximately 2-4 weeks after consenting

SECONDARY OUTCOMES:
Number of completed post-video questionnaires | Approximately 2-4 weeks after recording video

CONTACTS AND LOCATIONS:
Overall Officials: Paul Mueller, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials